CLINICAL TRIAL: NCT06130839
Title: Effects of Perturbation Based Training and Bobath-Based Trunk Exercises on Gait, Postural Control and Mobility in Post Stroke Patients
Brief Title: Perturbation Based Training And Bobath-Based Trunk Exercises On Gait , Postural Control And Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0245Saba Sheikh
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will be kept blinded about the intervention which the patients will be going to recieve.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perturbation based training (Experimental): 1. Stretching of the erector spinae,
  2. latissimus dorsi, gluteus Medius, gluteus minimums, and gluteus maximus (knee to chest) Pelvic Bridging Exercises
  3. Strengthening Exercises of latissimus dorsi muscle
  4. Pelvic Bridging Exercises include the gluteus maximus and quadriceps
  5. Rocker board:
  Trunk control exercises on Rocker Board in standing position first in medio-lateral direction for 10 min and then in anterio-posterior direction for 10 min with breaks in between.
  Interventions: Other: Rocker board training
- bobath based training (Experimental): 1. Stretching of the latissimus dorsi muscle
  2. Functional use and strengthening of the latissimus dorsi.
  3. Functional strengthening of abdominal and oblique abdominal muscles
  4. Placing exercises to facilitate trunk extension
  5. Rotations and counter-rotations (right and left) of the hips with the trunk extended Training of lumbar spine stabilizers
  Functional reach of shoulder, anterior, right, and left sides.
  Interventions: Other: Stable surface training

INTERVENTIONS:
Other: Rocker board training — Then intervention will be applied to the perturbation group as mention below at Rocker board (50 x 45 cm).the group will perform 36 sessions (4 times per week over 8 weeks) and effects of interventions will be measured before treatment, at 4th and after8th week (pre, mid and post intervention). Trunk control exercises on Rocker Board in standing position first in medio-lateral direction for 10 min and then in anterio-posterior direction for 10 min with breaks in between.
  Other Names: Experimental group
  Arms: perturbation based training
Other: Stable surface training — the group will perform 36 sessions (4 times per week over 8 weeks) and effects of interventions will be measured before treatment, at 4th and after 8th week (pre, mid and post intervention).
  Other Names: Experimental group
  Arms: bobath based training

SUMMARY:
This study compares two approaches for rehabilitating stroke patients: Perturbation-Based Training and Bobath-Based Trunk Exercises. The perturbation based training focuses on challenging patients with unexpected movements to improve their balance and stability. While the Bobath method, concentrating on facilitating normal movement patterns. The study aims to determine which approach yields better outcomes in terms of trunk control, balance, and functional recovery for stroke patients. This study will also enable the individual to be more independent and minimize their falls.

DETAILED DESCRIPTION:
Cerebrovascular is a leading cause of physical impairment and long-term disability in the globe. The complication of stroke is mobility impairment like balance, gait, and posture disorders. This impairment leads to a higher risk of falls, reduced ability in daily activities, and difficulty restoring the overall health and quality of life. Cerebrovascular accident is the second cause of fatality. Hence, one of the primary objectives in stroke rehabilitation is to restore postural stability and functional balance, which is a combination of dynamic, static and reactive balance. For improving postural stability and balance one such technique is the utilization of a rocker board, where a platform positioned on an unstable surface is used to challenge balance. Whilst rocker boards have been used effectively for, postural stability, injury prevention, rehabilitation and balance enhancement. Improvements in rocker board performance may be attributable to one or more of the following: muscle strengthening, enhanced intersegmental coordination, increase in brain activity in the supplementary motor area and/or enhanced feed-forward and feed-backward postural control mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk with or without ambulatory aids
* Able to follow commands.
* Patients in the subacute and chronic stages associated with stroke hemiparesis (time since
* stroke onset 6 months- 1 year)
* Scoring > 21 on MMSE

Exclusion Criteria:

* Patients who have severe limitations in passive range of motion at lower extremities
* Visual and sensory deficits
* Patient who has contracture
* Orthopedic or any other neurological disorder which impair balance.
* Patients undergoing any other balance training protocol.
* Patients with recurrent strokes
* Participants who are currently participating in another clinical trial or research study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale | 6 weeks
  It is used to measure motor impairment of the trunk after stroke. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance "Change will be measured from Baseline to 6 weeks"
Timed Up and Go Test | 6 weeks
  It is for the assessment of lower extremity function, mobility and fall risk. scoring criteria < 10 seconds = normal. < 20 seconds = good mobility; can walk outside alone; does not require a walking aid. < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid. "Change will be measured from Baseline to 6 weeks"
Postural Assessment Scale for Stroke Patient | 6 weeks
  It is used for the assessments of postural control in stroke patients. It measures the ability of an individual with stroke to maintain stable postures and equilibrium during positional changes. It consists of a 4-point scale where the items are scored from 0 to 3, and the total scoring ranges from 0 to 36. "Change will be measured from Baseline to 6 weeks"
Functional Gait Assessment | 6 weeks
  It is for assessment of postural stability during walk. 3 Normal is able to ambulate for 10 steps heel to toe with no staggering. 2 Mild impairment, ambulates 7-9 steps. 1 Moderate impairment, ambulates 4-7 steps. 0 Severe impairment, ambulates less than 4 steps heel to toe or cannot perform without assistance. "Change will be measured from Baseline to 6 weeks"

SECONDARY OUTCOMES:
Stroke Self-Efficacy Questionnaire | 6 weeks
  It evaluate self-efficacy as a result of being able to successfully perform a specific action in stroke patients. It is a self-reported questionnaire about level of confidence reported on a 0 to 10 scale (0 = not confident, 10 = very confident) when completing 13 activities of daily life following stroke. "Change will be measured from Baseline to 6 weeks"

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University Pakistan
Locations (1):
- LGH, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No